CLINICAL TRIAL: NCT00001313
Title: Evaluation of Patients With Known or Suspected Heart Disease (Screening Protocol)
Brief Title: Evaluation of Patients With Known or Suspected Heart Disease
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 920189; 92-H-0189
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-01-06

CONDITIONS: Peripheral Artery Disease; Coronary Disease; Diabetes and Heart Failure; Dilated Cardiomyopathy; Heart Failure; Renal Artery Stenosis; Pulmonary Hypertension
Keywords: Cardiac Diagnosis; Chest Pain; Hypertrophic Cardiomyopathy; Coronary Artery Disease; Microvascular Angina; Cardiac Investigation; Follow-up; Heart Disease
MeSH Terms: conditions — Peripheral Arterial Disease; Coronary Disease; Diabetes Mellitus; Heart Failure; Cardiomyopathy, Dilated; Renal Artery Obstruction; Hypertension, Pulmonary; Chest Pain; Cardiomyopathy, Hypertrophic; Coronary Artery Disease; Microvascular Angina; Heart Diseases

SUMMARY:
In this study researchers will admit and evaluate patients with known or suspected heart disease referred to the Cardiology Branch of the National Heart, Lung, and Blood Institute (NHLBI).

Patients participating in this study will undergo a general medical evaluation, including blood tests, urine, examination, chest x-ray and electrocardiogram (EKG). In addition, patients may be asked to have an echocardiogram (ultrasound scan of the heart) and to perform an exercise stress test.

These tests are designed to assess the types and causes of patient's heart diseases and to determine if they can participate in other, specific research studies.

DETAILED DESCRIPTION:
The principal mission of the NIH is the conduct of research that elucidates biological mechanisms, pathogenesis, and treatment of disease. Patients with known or suspected cardiovascular diseases are referred to NHLBI cardiologists for consideration of participation in clinical research protocols. However, eligibility for participation is often uncertain from referral information or even after an outpatient evaluation. The purpose of this protocol is to permit inpatient evaluation of patients for whom participation in clinical research protocols is under consideration in order to determine protocol eligibility by means of conventional laboratory and cardiovascular testing.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following is a representative list of the types of patient presentations and potential diagnoses eligible for this protocol:

1. Coronary artery disease with angina or inducible myocardial ischemia as determined by noninvasive testing.
2. Cardiomyopathies including congestive phenotypes.
3. Peripheral artery disease with intermittent claudication or limb-threatening ischemia.
4. Renovascular disease with uncontrolled hypertension, intermittent pulmonary edema, or evidence of ischemic nephropathy.
5. Upper extremity peripheral artery disease.
6. Diabetes with heart failure.
7. Pulmonary hypertension.

EXCLUSION CRITERIA:

Pregnancy, for those patients who require catheterization-based diagnostics.

Inability to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-05-10; Study Completion 2009-01-06

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Suburban Hospital, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland